CLINICAL TRIAL: NCT01697527
Title: Adoptive Transfer of NY-ESO-1 TCR Engineered Peripheral Blood Mononuclear Cells (PBMC) After a Nonmyeloablative Conditioning Regimen, With Administration of NY-ESO-1157-165 Pulsed Dendritic Cells and Interleukin-2, in Patients With Advanced Malignancies
Brief Title: Gene and Vaccine Therapy in Treating Patients With Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-000153; NCI-2012-01548 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — aldesleukin; Interleukin-2; fludarabine phosphate; Cyclophosphamide; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gene and vaccine therapy) (Experimental): CONDITIONING: Patients receive cyclophosphamide IV over 1 hour on days -5 to -4 and fludarabine phosphate IV over 30 minutes on days -4 to -1.
  TRANSPLANT: Patients receive NY-ESO-1 reactive TCR retroviral vector transduced autologous PBL IV on day 0. Patients also receive NY-ESO-1 (157-165) peptide pulsed dendritic cell vaccine therapy ID on days 1, 14, and 30 and aldesleukin SC BID on days 1-14. Patients may receive 3 additional doses of NY-ESO-1 (157-165) peptide pulsed dendritic cell vaccine therapy after day 90.
  Interventions: Biological: aldesleukin; Drug: fludarabine phosphate; Drug: cyclophosphamide; Other: laboratory biomarker analysis; Biological: NY-ESO-1 reactive TCR retroviral vector transduced autologous PBL; Biological: dendritic cell vaccine therapy; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography

INTERVENTIONS:
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Other: laboratory biomarker analysis — Correlative studies
Biological: NY-ESO-1 reactive TCR retroviral vector transduced autologous PBL — Undergo NY-ESO-1 reactive TCR retroviral vector transduced autologous PBL
  Other Names: anti-NY-ESO-1 TCR gene-engineered lymphocytes; anti-NY-ESO-1 TCR retroviral vector-transduced lymphocytes
Biological: dendritic cell vaccine therapy — Given NY-ESO-1-157-165 peptide pulsed dendritic cell vaccine ID
Radiation: fludeoxyglucose F 18 — Undergo PET scan using [18F] FDG tracer
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo fludeoxyglucose F18 PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
This phase II trial will examine whether genetically reprogramming a patient's disease fighting white blood cells may build an immune response to kill cancer cells that express the NY-ESO-1 protein. In this study, this genetic therapy will be given during a stem cell transplant along with a vaccine therapy. The vaccine will be made using the NY-ESO-1 protein and may help to stimulate the engineered immune response to tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether we can safely administer NY-ESO-1 T cell receptor transduced autologous peripheral blood mononuclear cells (PBMCs) (up to 1x10^9 cells) along with an NY-ESO-1 dendritic cell vaccine and low dose IL-2 to patients with advanced malignancies.

II. To evaluate the feasibility of delivering two patient-specific cell therapies, the NY-ESO-1 TCR transgenic peripheral blood mononuclear cell (PBMC) and NY-ESO-1 (157-165) peptide pulsed dendritic cells (DC), within a technically challenging study design that requires other significant interventions, like a lymphodepleting conditioning regimen and post-infusion of subcutaneous low dose interleukin (IL)-2 (aldesleukin).

III. To determine the rate of objective tumor responses, by Response Evaluation Criteria in Solid Tumors (RECIST) objective response criteria.

SECONDARY OBJECTIVES:

I. To determine the persistence of NY-ESO-1 TCR-engineered cells. This will be determined by temporally analyzing peripheral blood samples for the presence of T cells with the transduced NY-ESO-1 TCR by tetramer or dextramer analysis.

II. To explore the homing and persistence of the adoptively transferred NY-ESO-1 TCR-engineered PBMC in secondary lymphoid organs and tumor deposits via positron emission tomography (PET)-based imaging using the PET tracer fluorodeoxyglucose ([18F]FDG).

OUTLINE:

CONDITIONING: Patients receive cyclophosphamide intravenously (IV) over 1 hour on days -5 to -4 and fludarabine phosphate IV over 30 minutes on days -4 to -1.

TRANSPLANT: Patients receive NY-ESO-1 TCR transduced autologous PBMC IV on day 0. Patients also receive NY-ESO-1 (157-165) peptide pulsed dendritic cell vaccine therapy intradermally (ID) on days 1, 14, and 30 and aldesleukin subcutaneously (SC) twice daily (BID) on days 1-14. Patients may receive 3 additional doses of NY-ESO-1 (157-165) peptide pulsed dendritic cell vaccine therapy after day 90.

After completion of study treatment, patients are followed up at 30, 45, 60, and 75 days; every 3 months for 2 years; every 6 months for 3 years; and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or locally advanced cancers for which no alternative therapies with proven survival advantage are available.
* At least 1 lesion amenable for an outpatient biopsy; this should be a cutaneous or palpable metastatic site or a deeper site accessible by image-guided biopsy that is deemed safe to access by the treating physicians and interventional radiologists. Patients without accessible lesions for biopsy but with prior tissue available from metastatic disease would be eligible at the investigator's discretion.
* NY-ESO-1 positive malignancy by IHC utilizing commonly available NY-ESO-1 antibodies.
* HLA-A*0201 (HLA-A2.1) positivity by molecular subtyping.
* Age greater than or equal to 16 years old.
* Life expectancy greater than 3 months assessed by a study physician.
* A minimum of one measurable lesion defined as:

  a. Meeting the criteria for measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST).
* For patients with skin metastases, lesions selected as non-completely biopsied target lesion(s) that can be accurately measured and recorded by color photography with a ruler to document the size of the target lesion(s).
* No restriction based on prior treatments.
* ECOG performance status (PS) 0 or 1.
* Adequate bone marrow and hepatic function determined within 30-60 days prior to enrollment, defined as:

  1. Absolute neutrophil count > or = 1.5 x 109 cells/L.
  2. Platelets > or = 100 x 109/L.
  3. Hemoglobin > or = 10 g/dL.
  4. Aspartate and alanine aminotransferases (AST, ALT) < or = 2.5 x ULN (< or = 5 x ULN, if documented liver metastases are present).
  5. Total bilirubin < or = 2 x ULN (except patients with documented Gilbert's syndrome).
  6. Creatinine < 2 mg/dl (or a glomerular filtration rate > 60 mL/min).
* Must be willing and able to accept at least two leukapheresis procedures.
* Must be willing and able to accept at least two tumor biopsies.
* Must be willing and able to provide written informed consent.

Exclusion Criteria

* Previously known hypersensitivity to any of the agents used in this study.
* Received systemic treatment for cancer, including immunotherapy, within one month prior to initiation of dosing within this protocol. However, cell harvesting by leukapheresis may be performed before one month from prior therapy if the study investigators consider that it will not have a detrimental impact on the generation of the two cell therapies in this protocol.
* History of, or significant evidence of risk for, chronic inflammatory or autoimmune disease (eg, Addison's disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, inflammatory bowel disease, psoriasis, rheumatoid arthritis, systemic lupus erythematosus, hypophysitis, pituitary disorders, etc.). Patients will be eligible if prior autoimmune disease is not deemed to be active (e.x. fibrotic damage of the thyroid after thyroiditis or its treatment, with stable thyroid hormone replacement therapy). Vitiligo will not be a basis for exclusion.
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea or bleeding, or current acute colitis of any origin.
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 4 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed).
* HIV seropositivity or other congenital or acquired immune deficiency state, which would increase the risk of opportunistic infections and other complications during chemotherapy-induced lympho-depletion. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist.
* Hepatitis B or C seropositivity with evidence of ongoing liver damage, which would increase the likelihood of hepatic toxicities from the chemotherapy conditioning regimen and supportive treatments. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Clinically active brain metastases. Radiological documentation of absence of active brain metastases at screening is required for all patients. Prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment.
* Pregnancy or breast-feeding. Female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and 6 months after. All female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 14 days from starting the conditioning chemotherapy. The definition of effective contraception will be based on the judgment of the study investigators.
* Since IL-2 is administered following cell infusion:

  1. Patients will be excluded if they have a history of clinically significant ECG abnormalities, symptoms of cardiac ischemia or arrhythmias and have a left ventricular ejection fraction (LVEF) < 45% on a cardiac stress test (stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test)
  2. Similarly, patients who are 50 years old with a baseline LVEF < 45% will be excluded.
  3. Patients with ECG results of any conduction delays (PR interval >200ms, QTC > 480ms), sinus bradycardia (resting heart rate <50 beats per minute), sinus tachycardia (HR>120 beats per minute) will be evaluated by a cardiologist prior to starting the trial. Patients with any arrhythmias, including atrial fibrillation/atrila flutter, excessive ectopy (defined as >20 PVCs per minute), ventricular tachycardia, 3rd degree heart block will be excluded from the study unless cleared by a cardiologist.
  4. Patients with pulmonary function test abnormalities as evidenced by a FEV1/FVC< 70% of predicted for normality will be excluded.
* Received 3 or more prior myelotoxic treatment regimens.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2027-11-02 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Day +90
  Will be determined by RECIST 1.1 Criteria on Day +90

SECONDARY OUTCOMES:
NY-ESO-1 TCR transgenic cell persistence, quantitated in PBMC samples | Up to 6 years
NY-ESO-1 TCR transgenic cell tumor trafficking | Up to 40 days
  Regional uptake of fludeoxyglucose F18 within metastatic tumor sites and secondary lymphoid organs will be quantified by standardized uptake values (SUV) normalized to the body weight of the patient. The numbers of T lymphocytes will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ribas, MD, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- University of California at Los Angeles (UCLA ), Los Angeles, California, United States

REFERENCES:
- [Derived] Nowicki TS, Berent-Maoz B, Cheung-Lau G, Huang RR, Wang X, Tsoi J, Kaplan-Lefko P, Cabrera P, Tran J, Pang J, Macabali M, Garcilazo IP, Carretero IB, Kalbasi A, Cochran AJ, Grasso CS, Hu-Lieskovan S, Chmielowski B, Comin-Anduix B, Singh A, Ribas A. A Pilot Trial of the Combination of Transgenic NY-ESO-1-reactive Adoptive Cellular Therapy with Dendritic Cell Vaccination with or without Ipilimumab. Clin Cancer Res. 2019 Apr 1;25(7):2096-2108. doi: 10.1158/1078-0432.CCR-18-3496. Epub 2018 Dec 20. PMID 30573690